CLINICAL TRIAL: NCT02111187
Title: A Pharmacodynamic Pre-surgical Study of Hedgehog Pathway Inhibition With LDE225 in Men With High-risk Localized Prostate Cancer.
Brief Title: A Pre-surgical Study of LDE225 in Men With High-risk Localized Prostate Cancer
Acronym: LDE225
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J1402; NA_00091602 (Other: JHMIRB)
Record Dates: First submitted 2014-04-01; First posted 2014-04-11 (Estimated); Results first posted 2019-03-07 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2018-11

CONDITIONS: Prostate Cancer
Keywords: LDE225; High risk localized prostate cancer; Pre-surgical
MeSH Terms: conditions — Prostatic Neoplasms | interventions — sonidegib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LDE225 (Arm1) (Active Comparator): Treatment arm (Arm 1) will receive LDE225 by mouth 800 mg daily for 4 weeks (+/- 3 days)
  Interventions: Drug: LDE225
- Observation Arm (Arm2) (No Intervention): Observation Arm (Arm2) will receive no treatment prior to prostatectomy.

INTERVENTIONS:
Drug: LDE225 — Sonidegib was given as an oral drug at 800mg daily for 28 days prior to prostetoctomy
  Other Names: Sonidegib
  Arms: LDE225 (Arm1)

SUMMARY:
This trial is designed as a randomized two-arm (LDE225 vs. observation groups) open-label prospective clinical trial in men with localized high-risk prostate cancer undergoing radical prostatectomy.

The investigators propose to determine the effects of LDE225 on neoplastic prostate tissue from men at high risk of systemic disease progression, by comparing pre-surgical core-biopsy specimens to tumor tissue harvested at the time of prostatectomy.

DETAILED DESCRIPTION:
High-risk patients will be identified based on their core-needle biopsy features, PSA levels, and clinical stage. After obtaining baseline laboratory and clinical values (including an ECG, PSA, hematologic, and renal and hepatic panels), men will receive oral LDE225 800 mg/day or observation daily for 4 weeks (±3 days) prior to prostatectomy. Patients will have a clinical visit and an ECG and laboratory testing will be performed at 2 weeks and then again at 4 weeks, including a 4-week pre-prostatectomy measurement of PSA and a blood sample to determine plasma LDE225 levels. Men will undergo radical prostatectomy (with bilateral pelvic lymphadenectomy as appropriate), at which point two 250-mg biopsies of prostate tissue will be obtained, frozen and stored for analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to any screening procedures.
2. Age 18 years or older.
3. Histologically-documented prostatic adenocarcinoma in ≥2 cores
4. ECOG performance status ≤2
5. Localized prostate cancer with at least one of the following NCCN high-risk features:

   * Gleason sum ≥8
   * PSA >20 ng/mL
   * Clinical stage ≥T3
6. Must be a candidate for radical prostatectomy
7. No evidence of known metastatic disease (M0 or Mx allowed)
8. Adequate bone marrow, liver and renal function as specified below:

   * Absolute neutrophil count (ANC) ≥ 1500/µL
   * Hemoglobin (Hgb) ≥ 9.0 g/dL
   * Platelets ≥100,000/µL
   * Serum total bilirubin ≤ 1.5 x ULN (upper limit of normal)
   * AST and ALT ≤ 2.5 x ULN
   * Plasma creatine phosphokinase (CK) < 1.5 x ULN, if known
   * Serum creatinine ≤ 1.5 x ULN [or 24-hour creatinine clearance ≥ 50ml/min]
9. Patient is able to swallow and retain oral medications

Exclusion Criteria:

1. Patients who have had major surgery within 4 weeks of enrollment.
2. Patients with concurrent uncontrolled medical conditions that may interfere with their participation in the study.
3. Patients unable to take oral drugs (e.g. lack of physical integrity of the upper GI tract or known malabsorption syndromes).
4. Patients who have previously been treated with LDE225 or other Hh pathway inhibitors
5. Patients who have neuromuscular or muscular disorders (e.g. inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis and spinal muscular atrophy) or are on concomitant treatment with drugs that are known to cause rhabdomyolysis (such as statins and fibrates), and that cannot be discontinued at least 2 weeks prior to starting LDE225. If it is essential that the patient stays on a statin for hyperlipidemia, only pravastatin may be used with extra caution. Patients should not plan to embark on a new strenuous exercise regimen after initiation of study treatment. (NB: Muscular activities, such as strenuous exercise, that can result in significant increases in plasma CK levels should be avoided whilst on LDE225 treatment).
6. Patients who have taken part in an experimental drug study within 4 weeks or 5 half-lives (whichever is longer) of initiating treatment with LDE225.
7. Patients who are receiving other anti-neoplastic therapy (e.g. chemotherapy, targeted therapy or radiotherapy) concurrently or within 2 weeks of starting LDE225.
8. Patients taking moderate/strong inhibitors or inducers of CYP3A4/5 or drugs metabolized by CYP2B6 or CYP2C9 that have narrow therapeutic index, and that cannot be discontinued before starting treatment with LDE225. Medications that are strong CYP3A4/5 inhibitors should be discontinued for at least 7 days and strong CYP3A/5 inducers for at least 2 weeks prior to starting treatment with LDE225.
9. No concurrent use of statins (except for pravastatin, if absolutely necessary)
10. No concurrent warfarin or Coumadin-derivatives
11. Impaired cardiac function or significant heart disease, including any one of the following:

    * Angina pectoris within 3 months
    * Acute myocardial infarction within 3 months
    * QTc >450 msec on the screening ECG
    * A past medical history of clinically significant ECG abnormalities or a family history of prolonged QT-interval syndrome
    * Other clinically significant heart disease (e.g. heart failure, uncontrolled/labile hypertension, or history of poor compliance with an antihypertensive regimen)
12. Patients who are not willing to apply highly effective contraception during the study and through the duration of LDE225 treatment.

    * Male patients must use highly effective (double barrier) methods of contraception (e.g., spermicidal gel plus condom) for the entire duration of the study, and continuing using contraception and refrain from fathering a child for 6 months following the last dose of the study drug. A condom is also required to be used by vasectomized men as well as during intercourse with a male partner in order to prevent delivery of the study treatment via seminal fluid. Sexually active males must be willing to use a condom during intercourse while taking the study drug and for 6 months after stopping investigational medications and agree not to father a child during this period.
13. Patients unwilling or unable to comply with the research protocol.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-01-18 (Actual); Study Completion 2017-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Antonarakis, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- LDE225 (Arm1): Treatment arm (Arm 1) will receive LDE225 by mouth 800 mg daily for 4 weeks (+/- 3 days)
  LDE225
Period: Overall Study
Arm/Group | LDE225 (Arm1) | Observation Arm (Arm2)
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LDE225 (Arm1) | Observation Arm (Arm2) | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 7 | 7 | 14
Race/Ethnicity, Customized [Number; unit: participants]
  caucasian | 7 | 6 | 14
  African-American | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Tissue Gli1 Expression Levels Using qRT-PCR Analysis in Each Group (LDE225 and Observation)
Description: This was defined as the number of patients who achieved at least a two-fold reduction in GLI1 expression in post-treatment vs. pre-treatment tumor tissues.
Time Frame: Up to 3 Years
Measure: Count of Participants; unit: Participants
Arm/Group | LDE225 (Arm1) | Observation Arm (Arm2)
Number analyzed (Participants) | 7 | 7
Participants | 6 | 0

2. Secondary Outcome: Percentage of Participants With a Pathological Effect of Presurgical Treatment With LDE225
Description: To determine whether presurgical treatment with LDE225 can exert a pathological effect on high-risk tumors (i.e. increase apoptosis, decrease proliferation).
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | LDE225 (Arm1) | Observation Arm (Arm2)
Number analyzed (Participants) | 7 | 7
Participants
  Pathologic Gleason Sum 7 | 1 | 1
  Pathologic Gleason Sum 9 | 5 | 6
  Pathologic Gleason Sum 10 | 1 | 0

3. Secondary Outcome: Effect of LDE225 on PSA Recurrence Following Prostatectomy
Description: To evaluate whether presurgical treatment with LDE225 diminishes the risk of PSA recurrence following prostatectomy.
Time Frame: Up to 3 years
Measure: Median (Full Range); unit: ng/ml
Arm/Group | LDE225 (Arm1) | Observation Arm (Arm2)
Number analyzed (Participants) | 7 | 7
ng/ml | 12.0 [3.2 to 29.7] | 7.4 [2.4 to 10.4]

4. Secondary Outcome: Number of Participants With Adverse Events in Each Group (LDE225 and Observation)
Description: Safety and tolerability, including any drug-related toxicities of Sonidegib, were reported via CTCAE version 4.0.
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | LDE225 (Arm1) | Observation Arm (Arm2)
Number analyzed (Participants) | 7 | 7
Participants | 3 | 0

ADVERSE EVENTS:
Time Frame: 1 year and 6 months
Arm/Group | LDE225 (Arm1) | Observation Arm (Arm2)
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 3/7 | 0/7
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LDE225 (Arm1) (N=7) | Observation Arm (Arm2) (N=7)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Increased CK level (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
AST/ALT elevated (Hepatobiliary disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Dry mouth (Endocrine disorders) | 1 (1) | 0 (0)
arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
dysgeusia (Endocrine disorders) | 1 (1) | 0 (0)
myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-06): https://cdn.clinicaltrials.gov/large-docs/87/NCT02111187/Prot_SAP_000.pdf